CLINICAL TRIAL: NCT05144503
Title: A Safety and Performance Assessment of the SpherePVI™ Catheter and the Affera Mapping and Ablation System to Treat Paroxysmal Atrial Fibrillation
Brief Title: Safety and Performance of the SpherePVI™ Catheter to Treat Paroxysmal Atrial Fibrillation
Acronym: SpherePVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00012
Record Dates: First submitted 2021-10-20; First posted 2021-12-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SpherePVI™ Catheter (Experimental): Subjects treated with the SpherePVI™ Catheter
  Interventions: Device: SpherePVI™ Catheter

INTERVENTIONS:
Device: SpherePVI™ Catheter — SpherePVI™ Catheter with the Affera Mapping and Ablation System

SUMMARY:
A prospective, single-arm, single-center study to evaluate the safety, performance, and effectiveness of the SpherePVI™ Catheter for treating paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic paroxysmal atrial fibrillation (PAF) documented by:

   * A physician's note indicating recurrent, self-terminating AF
   * At least two electrocardiographically documented AF episodes within 12 months prior to enrollment
2. Failure or intolerance of at least one Class I-IV anti-arrhythmic drug.
3. Suitable candidate for catheter ablation.
4. Age ≥ 18 and < 75 years.
5. Able and willing to give informed consent.
6. Able and willing, and has ample means to comply with all pre-procedure, post-procedure and follow-up testing requirements

Exclusion Criteria:

1. Continuous AF lasting more than 7 days.
2. AF secondary to electrolyte imbalance, thyroid disease, acute alcohol intoxication, or reversible or non-cardiac cause.
3. Previous left atrial catheter or surgical ablation (including septal closure or left atrial appendage closure).
4. Valvular cardiac surgical/percutaneous procedure (e.g., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve).
5. Any carotid stenting or endarterectomy.
6. Any cardiac procedure (surgical or percutaneous) or percutaneous coronary intervention within 90 days prior to the initial procedure.
7. Coronary artery bypass graft (CABG) procedure within the 6 months prior to the index ablation procedure.
8. Awaiting cardiac transplantation or other cardiac surgery within 12 months following the initial ablation procedure.
9. Presence of any type of implantable cardiac defibrillator (with or without biventricular pacing function).
10. Documented thromboembolic event (stroke or transient ischemic attack) within the past 6 months (180 days).
11. Documented left atrial thrombus on imaging.
12. History of blood clotting or bleeding abnormalities.
13. Any condition contraindicating chronic anticoagulation.
14. Myocardial infarction (MI) within the 3 months (90 days) prior to the initial procedure.
15. Body mass index >40 kg/m2.
16. Left atrial diameter >50 mm (anteroposterior).
17. Diagnosed atrial myxoma.
18. Left ventricular ejection fraction (EF) < 40%.
19. Uncontrolled heart failure or NYHA Class III or IV heart failure.
20. Rheumatic heart disease.
21. Hypertrophic cardiomyopathy.
22. Unstable angina.
23. Moderate to severe mitral valve stenosis.
24. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2)
25. Primary pulmonary hypertension.
26. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition.
27. Renal failure requiring dialysis.
28. Acute illness, active systemic infection, or sepsis.
29. Significant congenital anomaly or medical problem that, in the opinion of the investigator, would preclude enrollment in this study or compliance with follow-up requirements or would impact the scientific soundness of the clinical trial results.
30. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence.
31. Current or anticipated participation in any other clinical trial of a drug, device, or biologic during the duration of the study, unless pre-approved by the Sponsor.
32. Presence of intramural thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation.
33. Known drug or alcohol dependency.
34. Life expectancy less than 12 months.
35. Vulnerable subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects experiencing a primary safety event | Up to 6 months
  The primary safety outcome is the incidence of the following serious device-related Primary Adverse Events (AEs):
  * Death (within 7 days)
  * Myocardial infarction (within 7 days)
  * Persistent phrenic nerve palsy (within 7 days)
  * Transient ischemic attack (TIA) (within 7 days)
  * Stroke/cerebrovascular accident (CVA) (within 7 days)
  * Thromboembolism (within 7 days)
  * Major vascular access complications / bleeding (within 7 days)
  * Heart block (within 7 days)
  * Gastroparesis (within 7 days)
  * Severe pericarditis (within 7 days)
  * Pulmonary edema (within 7 days)
  * Hospitalization (initial and prolonged) due to cardiovascular or pulmonary AE (within 7 days)
  * Cardiac tamponade / perforation (within 30 days)
  * Pulmonary vein stenosis (within 180 days)
  * Atrio-esophageal fistula (within 180 days)
Percentage of subjects with acute procedure success | During Procedure
  The primary efficacy outcome is acute electrical isolation of all pulmonary veins using the study device

SECONDARY OUTCOMES:
Percentage of subjects experiencing a device- or procedure-related SAE | 12 months
  The secondary safety outcome is the incidence of device- or procedure-related SAEs as assessed at each follow-up visit.
Product performance evaluated on a 5-point semi-quantitative scale ("strongly disagree" to "strongly agree") | During Procedure
  Acute product performance will be evaluated during the procedure and includes the following:
  * SpherePVI™ Catheter handling sufficient to reach reasonable intended targets, as determined by the physician:
    * catheter delivery to the desired ablation sites
    * completion of ablation procedure
    * safe removal of catheter from the subject
  * Electroanatomical navigation and/or mapping sufficient to aid the procedure (if used)
  * Generation of acceptable acute ablation lesions
Percentage of subjects free from documented recurrence outside of the blanking period | 12 months
  Chronic efficacy will be evaluated as freedom from documented arrhythmia recurrence outside of a 90-day blanking period. Failure will be reported as both (i) recurrence of AF and (ii) recurrence of any atrial tachyarrhythmia (AF, atrial tachycardia, or atrial flutter).
Percentage of pulmonary veins remaining isolated at remapping | 75 days
  Chronic efficacy evaluated as the number of pulmonary veins that remain isolated during an optional remapping procedure as
Percentage of patients with all pulmonary veins isolated at remapping | 75 days
  Chronic efficacy evaluated as the number of patients with all pulmonary veins isolated during an optional remapping procedure as

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy VY, Peichl P, Kautzner J, Anter E, Metzner A, Koruth J, Jais P, Rackauskas G, Petru J, Funasako M, Marinskis G, Turagam M, Aidietis A, Selma JM, Nejedlo V, Kueffer F, Tarakji KG, Natale A, Neuzil P. One-year outcomes of a conformable single-shot pulsed-field ablation catheter for the treatment of paroxysmal atrial fibrillation. Heart Rhythm. 2025 Oct;22(10):2551-2561. doi: 10.1016/j.hrthm.2025.04.031. Epub 2025 Apr 26. PMID 40294729
- [Background] Reddy VY, Anter E, Peichl P, Rackauskas G, Petru J, Funasako M, Koruth JS, Marinskis G, Turagam M, Aidietis A, Kautzner J, Natale A, Neuzil P. First-in-human clinical series of a novel conformable large-lattice pulsed field ablation catheter for pulmonary vein isolation. Europace. 2024 Mar 30;26(4):euae090. doi: 10.1093/europace/euae090. PMID 38584468